CLINICAL TRIAL: NCT07307612
Title: Improving Lung Health in Premature Babies Through Early Nutrition: The More & Early Nutritional Delivery for Bronchopulmonary Dysplasia (MEND-BPD) Trial
Brief Title: High-energy Human Milk Diets in the First Two Weeks After Birth to Reduce BPD in Extremely Preterm Infants
Acronym: MEND-BPD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ariel A. Salas, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-300016002
Record Dates: First submitted 2025-12-24; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Extreme Prematurity; Enteral Nutrition; Bronchopulmonary Dysplasia
Keywords: Prematurity; Extreme
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Following written informed consent, participants are assigned in a 2:1 ratio to either the intervention (supplementation) or control (standard diet) group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain trial integrity, nutrition room staff that are independent of clinical care will prepare the feeding syringes without DHA/ARA labels to ensure clinicians, parents, and evaluators remain masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-energy Group (Active Comparator): The intervention group receives a standard fortified human milk (maternal or donor) diet plus the DHA/ARA supplement for the first 14 days. Infants in this group will be secondarily assigned to either a low-dose (60/120 mg/kg/day) or high-dose (120/240 mg/kg/day) DHA/ARA supplement.
  Interventions: Dietary Supplement: High-energy group
- Standard-energy Group (Other): The control group receives a standard fortified human milk (maternal or donor) diet for the first 14 days.
  Interventions: Other: Standard-energy group

INTERVENTIONS:
Dietary Supplement: High-energy group — Study participants assigned to the intervention group will receive a standard, fortified human milk diet plus a DHA/ARA supplement during the first 2 weeks after birth.
  Arms: High-energy Group
Other: Standard-energy group — Study participants assigned to the intervention group will receive a standard, fortified human milk diet during the first 2 weeks after birth.
  Arms: Standard-energy Group

SUMMARY:
This Phase II, parallel-group, masked, randomized clinical trial aims to evaluate whether a DHA/ARA-enriched, fortified human milk diet administered during the first 14 days of life reduces respiratory morbidity and improves lung function in extremely preterm (EPT) infants (born at ≤28 weeks gestation).

DETAILED DESCRIPTION:
This is a masked randomized clinical trial in which extremely preterm infants fed human milk will be randomly assigned to receive either a docosahexaenoic acid/arachidonic acid (DHA/ARA)-enriched, fortified human milk diet (intervention group) or a standard fortified human milk diet (control group) during the first 14 days after birth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 28 weeks of gestation
* Postnatal age < 72 hours

Exclusion Criteria:

* Congenital malformations
* Chromosomal anomalies
* Terminal illness needing to limit or withhold support

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-05-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Severity of respiratory morbidity | 0 - 120 days
  A scoring system that defines severity of respiratory morbidity (bronchopulmonary dysplasia severity) based on the amount of ventilatory support and the need for supplemental oxygen at 36 weeks postmenstrual age using the Jensen criteria, an ordinal scale ranging from 0 (no respiratory support) to 1 (mild BPD: low-flow nasal cannula ≤2 L/min requirement); 2 (moderate BPD: non-invasive respiratory support, including high-flow nasal cannula >2 L/min, CPAP, or non-invasive positive pressure ventilation); 3 (severe BPD - invasive mechanical ventilation); or 4 (death), with progressively higher scores indicating increasing respiratory morbidity and worse clinical outcomes.
Non-invasive impulse oscillometry measurements of pulmonary mechanics | 40 - 120 days
  Using the N-100 Neo Oscillometry device, we will determine the area under the reactance curve (AX)

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | 40 - 120 days
  Defined as the need for ventilatory support or supplemental oxygen at 36 weeks of postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States